CLINICAL TRIAL: NCT02976870
Title: Hydronephrosis After Anterior Lumbar Interbody Fusion (ALIF)
Acronym: HAALIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12SP006
Record Dates: First submitted 2012-10-05; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Hydronephrosis
Keywords: Hydronephrosis; Anterior Lumbar Interbody Fusion
MeSH Terms: conditions — Hydronephrosis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasound (Experimental): Single ultrasound scan of kidney on side of body where ALIF was performed. If hydronephrosis of this kidney is detected, the second kidney will also be scanned.
  Interventions: Radiation: Ultrasound

INTERVENTIONS:
Radiation: Ultrasound — Single ultrasound scan of kidney on side of body where ALIF was performed. If hydronephrosis of this kidney is detected, the second kidney will also be scanned.

SUMMARY:
Anterior lumbar spinal surgery involves making an incision through the abdomen of the patient in order to access the spine. During this process, several internal structures are pushed aside in order to gain access. One of these structures is the ureter, whose function is to drain urine from the kidney to the bladder. One potential complication that can arise from this is dilation of the kidney - known as hydronephrosis. The aim of this study is to identify whether hydronephrosis after Anterior Lumbar Interbody Fusion (ALIF) is complication, in order to bring this to the attention of health care professionals when considering this kind of surgery.

DETAILED DESCRIPTION:
A total of 40 patients who have had ALIF surgery will be invited to have an ultrasound scan of their kidney on the side where the operation was performed (where the scar is). Should hydronephrosis of this kidney be detected, the investigators will go on to scan the second kidney. Should hydronephrosis be detected the patient will be given a letter to take to their General Practitioner (GP) advising them to be referred to a Urologist.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Has the mental capacity to provide informed consent for participation within the study
* Patients who have had anterior lumbar spinal surgery at least 12 months ago and no longer than 5 years ago

Exclusion Criteria:

* Unable to understand written or verbal information regarding the study
* Multiple abdominal surgeries prior to spinal surgery
* Previous renal complication such as renal strictures or hydronephrosis/use of stents
* Pregnancy
* Structural anomalies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Identification of hydronephrosis on ultrasound scan | 12 month
  Each participant will have an ultrasound scan of their kidney. After this ultrasound scan participant will have no further involvement in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Bronek Boszczyk, PD. Dr.med., Principal Investigator — The Centre for Spinal Studies and Surgery, Queen's Medical Centre, Nottingham, NG7 2UH.
Locations (1):
- Queen's Medical Centre, Nottingham, United Kingdom